CLINICAL TRIAL: NCT04906109
Title: A Randomized, Open-label, Single-dose, 2x2 Crossover Study to Compare the Safety/Tolerability and Pharmacokinetics Between and DA-2803 and Vemlidy® After Meal in Healthy Adults
Brief Title: Clinical Study to Evaluate the Pharmacokinetics, Safety and Tolerability of DA-2803 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA2803_BE_I
Record Dates: First submitted 2021-05-24; First posted 2021-05-28 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-06

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference-Test (Experimental)
  Interventions: Drug: Vemlidy Tab; Drug: DA-2803 Tab
- Test-Reference (Experimental)
  Interventions: Drug: Vemlidy Tab; Drug: DA-2803 Tab

INTERVENTIONS:
Drug: Vemlidy Tab — 1T
  Other Names: Reference
Drug: DA-2803 Tab — 1T
  Other Names: Test

SUMMARY:
This study is an open-label, randomized, single dose, crossover study to evaluate the pharmacokinetics, safety and tolerability of DA-2803 in healthy subjects

DETAILED DESCRIPTION:
To healthy subjects of ninety-six (96), following treatments are administered dosing in each period and wash-out period is a minimum of 14 days.

Reference drug: Vemlidy Tab. / Test drug: DA-2803 Tab. Pharmacokinetic blood samples are collected up to 72hrs. The pharmacokinetic characteristics and safety are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, aged between ≥ 19 and ≤ 45 years old at the time of screening.
* Calculated body mass index (BMI) of ≥ 18.0 and ≤ 28.0 kg/m2

  * BMI = Weight(kg)/ Height(m)2
* Individuals who agreed proper contraception during the study and did consent to not donation of sperm and ovum before the termination of study
* Individuals who voluntary decide to participate and agrees in writing to comply with the precautions after hearing and fully understanding the detailed explanation of this clinical trial

Exclusion Criteria:

* History or presence of clinically significant and sever active cardiovascular, respiratory, hepatobiliary, renal, hematological, gastrointestinal, endocrine, immune, dermatologic, neurologic, or psychiatric disorder.
* Any medical history that may affect drug absorption, distribution, metabolism and excretion.
* Individuals who had history of hypersensitivity to Investigational drugs, derivative drugs or others drugs(aspirin and antibiotics etc.)
* Any clinically significant chronic medical illness.
* Any genetic disease including galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
* Individuals with one of the following laboratory test results in screening.

  * AST, ALT > UNL (upper normal limit) x 1.5
  * Creatinine clearance ≤ 60 mL/min
  * Positive test results at HBs Ag, anti-HCV Ab, anti-HIV Ab, VDRL.
* Use of any prescription drugs and herbal preparations within 14 days prior to study drug administration and use of over-the-counter medications within 10 days prior to study drug administration.
* Individuals who cannot eat standard meal provided from clinical trial center.
* Donation of blood within 60 days prior to study drug administration or apheresis within 30 days prior to the first IP administration.
* Individuals who had received a blood transfusion within 60 days prior to study drug administration.
* Exposure to any investigational drug within 6 months prior to the first IP administration.
* Individuals taking any drugs inducing or inhibiting drug metabolizing enzymes including barbiturates within 30 days prior to the first IP administration.
* Individuals who had drinking (alcohol > 21unit/week) within 14 days prior to screening.
* Heavy smoking (more than 10 cigarettes/day) within 14 days prior to screening.
* Subjects having been deemed inappropriate for the trial as determined by the investigator.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
AUCt of DA-2803, Vemlidy | pre-dose(0 hour), 0.08, 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72 hour
  Area under the DA-2803/Vemlidy concentration in blood-time curve from zero to final
Cmax of DA-2803, Vemlidy | pre-dose(0 hour), 0.08, 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72 hour
  The maximum DA-2803/Vemlidy concentration in blood sampling time t

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No